CLINICAL TRIAL: NCT05021341
Title: Bioavailability of Berberine and Dihydroberberine and Their Impact on Glycemia
Acronym: BBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lindenwood University (Other)
Collaborators: NNB Nutrition (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: IRB-20-173
Record Dates: First submitted 2021-07-01; First posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Glycemia
MeSH Terms: interventions — Berberine

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, crossover study design
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Berberine (Active Comparator): 500 mg of Berberine
  Interventions: Dietary Supplement: Berberine
- Dihydroberberine 200 (Active Comparator): 200 mg of Dihydroberberine
  Interventions: Dietary Supplement: Dihydroberberine 200
- Dihydroberberine 100 (Active Comparator): 100 mg of Dihydroberberine
  Interventions: Dietary Supplement: Dihydroberberine 100
- Placebo (Placebo Comparator): Maltodextrin
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Berberine — For each visit, all participants will report to the laboratory between 0600 - 1000 hours after observing an 8 - 10 hr fast. Participants will ingest the double-blinded supplement (500 mg of berberine) at specific times, the day before and morning of study visits 2 - 5. For each visit, participants will have their heart rate, blood pressure, body mass, and height measured. After final ingestion of their assigned supplementation dose, standard multiple sample phlebotomy approaches will be used to collect 10 mL of venous blood from a forearm vein at 0, 20, 40, 60, 90, and 120 minutes post-supplement ingestion. After donating baseline blood sample (0-min) a standard test meal, white bread, and glucose powder mixed in 250 mL of water. The complete nutritional breakdown of the test meal is anticipated to be 382 kcal, 3.2 grams of fat, 80.6 grams of carbohydrate, and 7.64 grams of protein.
  Arms: Berberine
Dietary Supplement: Dihydroberberine 200 — For each visit, all participants will report to the laboratory between 0600 - 1000 hours after observing an 8 - 10 hr fast. Participants will ingest the double-blinded supplement (200 mg of dihydroberberine) at specific times, the day before and morning of study visits 2 - 5. For each visit, participants will have their heart rate, blood pressure, body mass, and height measured. After final ingestion of their assigned supplementation dose, standard multiple sample phlebotomy approaches will be used to collect 10 mL of venous blood from a forearm vein at 0, 20, 40, 60, 90, and 120 minutes post-supplement ingestion. After donating baseline blood sample (0-min) a standard test meal, white bread, and glucose powder mixed in 250 mL of water. The complete nutritional breakdown of the test meal is anticipated to be 382 kcal, 3.2 grams of fat, 80.6 grams of carbohydrate, and 7.64 grams of protein.
  Arms: Dihydroberberine 200
Dietary Supplement: Dihydroberberine 100 — For each visit, all participants will report to the laboratory between 0600 - 1000 hours after observing an 8 - 10 hr fast. Participants will ingest the double-blinded supplement (100 mg of dihydroberberine) at specific times, the day before and morning of study visits 2 - 5. For each visit, participants will have their heart rate, blood pressure, body mass, and height measured. After final ingestion of their assigned supplementation dose, standard multiple sample phlebotomy approaches will be used to collect 10 mL of venous blood from a forearm vein at 0, 20, 40, 60, 90, and 120 minutes post-supplement ingestion. After donating baseline blood sample (0-min) a standard test meal, white bread and glucose powder mixed in 250 mL of water. The complete nutritional breakdown of the test meal is anticipated to be 382 kcal, 3.2 grams of fat, 80.6 grams of carbohydrate, and 7.64 grams of protein.
  Arms: Dihydroberberine 100
Dietary Supplement: Placebo — For each visit, all participants will report to the laboratory between 0600 - 1000 hours after observing an 8 - 10 hr fast. Participants will ingest the double-blinded supplement (Maltodextrin placebo) at specific times, the day before and morning of study visits 2 - 5. For each visit, participants will have their heart rate, blood pressure, body mass, and height measured. After final ingestion of their assigned supplementation dose, standard multiple sample phlebotomy approaches will be used to collect 10 mL of venous blood from a forearm vein at 0, 20, 40, 60, 90, and 120 minutes post-supplement ingestion. After donating baseline blood sample (0-min) a standard test meal, white bread, and glucose powder mixed in 250 mL of water. The complete nutritional breakdown of the test meal is anticipated to be 382 kcal, 3.2 grams of fat, 80.6 grams of carbohydrate, and 7.64 grams of protein.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the bioavailability of berberine and dihydroberberine and their impact on changes in plasma concentrations of glucose and insulin.

DETAILED DESCRIPTION:
Once determined eligible and provided consent, participants will be assigned in a randomized, double-blind, placebo-controlled, crossover fashion. Eligible study participants will complete one of four testing conditions. For each testing condition, study participants will arrive in the lab after observing an overnight fast. Upon arrival, participants will donate the first of six venous blood samples. Follow-up blood samples will be collected at 20, 40, 60, 90, and 120 minutes. All collected samples will be collected into two, 4mL EDTA tubes and have aliquots of 600 ul of plasma isolated and frozen at -80 degrees celsius. Collected plasma will be analyzed for changes in berberine, glucose, and insulin. Participants will observe a minimum of 72 hours washout between conditions

ELIGIBILITY:
Inclusion Criteria:

* All participants will be between the ages of 18-45 years.
* Participants will be healthy and free of disease as determined by evaluation of a medical history
* Body mass index (BMI) between 18.5 - 30 kg/m^2

Exclusion Criteria:

* Those individuals less than 18 and greater than 45 years of age will be excluded.
* Participants younger than 18 are excluded due to necessity of parental consent.
* Participants greater than 45 years old lie outside of the target demographic for the current study.
* As indicated on a medical history form they complete, any individual who is currently being treated for or diagnosed with any cardiac, respiratory, endocrine, psychiatric, musculoskeletal, renal, hepatic, neuromuscular or metabolic disease or disorder.
* Additional exclusion criteria include: participants with a fasting capillary blood glucose level > 100 mg/dL.
* Current smokers (including vaping) or have quit within the past six months.
* Any over-the-counter or prescription drugs and/or dietary supplements that are known or are purported to impact glycemia and insulinemia.
* Currently or have been following with the past 30 days a ketogenic or very-low carbohydrate diet.
* Participants who are determined to not be weight stable defined as measured body mass deviating by 2% or more.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2020-11-04 (Actual); Study Completion 2020-11-04 (Actual)

PRIMARY OUTCOMES:
Berberine | 30 days
  Changes in plasma berberine levels after supplementing 500 mg of berberine
Dihydroberberine 200 | 30 days
  Changes in plasma berberine levels after supplementing 200 mg of dihyrdoberberine
Dihydroberberine 100 | 30 days
  Changes in plasma berberine levels after supplementing 100 mg of dihyrdoberberine
Glucose | 30 days
  Changes in plasma glucose levels after supplementing either berberine or dihyrdoberberine
Insulin | 30 days
  Changes in insulin levels after supplementing either berberine or dihyrdoberberine

CONTACTS AND LOCATIONS:
Overall Officials: Chad Kerksick, PhD, Principal Investigator — Lindenwood University
Locations (1):
- Lindenwood University, Saint Charles, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Researchers do not plan to share data to other/outside researchers. Upon study completion, a manuscript will be developed and submitted for publication.